CLINICAL TRIAL: NCT02229734
Title: Fairly Brief Androgen Suppression and Stereotactic Radiotherapy for High Risk Prostate Cancer - Protocol 2
Acronym: FASTR-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Glenn Bauman, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FASTR-2
Record Dates: First submitted 2014-08-27; First posted 2014-09-01 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation plus Androgen Supression (Experimental): Radiation plus Androgen Suppression give as stereotactic radiation 7gray (Gy) per week x 5 weeks and leuprolide 45mg every 6 months for 18 months
  Interventions: Radiation: Radiation; Drug: Androgen Suppression

INTERVENTIONS:
Radiation: Radiation — Radiation: Radiotherapy 7 gray (Gy) per week over 5 weeks (35Gy)
Drug: Androgen Suppression — Leuprolide 45mg every 6 months for a total of 18 months
  Other Names: LHRH agonist

SUMMARY:
This study will explore the combination of a stereotactic body radiation therapy (SBRT) approach combined with one year of luteinizing hormone releasing hormone (LHRH) agonist for older men with high risk prostate cancer, or men unwilling to undertake conventionally fractionated therapy and three years of adjuvant hormone therapy.

The purpose of this study is to examine the safety of a shorter course of radiation treatment combined wtih androgen deprivation therapy.

DETAILED DESCRIPTION:
Randomized controlled trials have established the improved efficacy (better biochemical control and disease free survival) of combined radical radiation (70-80 Gy over 7-8 weeks) combined with long term hormone therapy (2-3 years of adjuvant LHRH agonist) compared to a primary hormone therapy or radiation therapy alone in men with locally advanced/high risk disease. While this approach may be tolerable in fit individuals, this combination may not be well tolerated by frail individuals, or those who live at a distance who may find it difficult to attend for 7 weeks of radiation treatments. Those individuals with co-morbidities such as diabetes, coronary artery disease or osteoporosis may have those conditions exacerbated by long term hormone therapy.

The combination of short course radiation and hormone therapy was explored in the FASTR trial. As part of the trial, patients received 12 months of hormone therapy with radiation treatment to the pelvic lymph nodes (dose of 25 Gy in 5 fractions, 1 fraction per week) concomitant with radiation treatment to the prostate (dose of 40 Gy in 5 fractions, 1 fraction per week). The study was discontinued due to toxicity. For the FASTR-2 study, these concerns are being addressed through the use of a lower total dose to the prostate (35 Gy in 5 fractions, 1 fraction per week). Given the uncertainty of the benefit of pelvic nodal radiation in prostate cancer, it was decided to omit the pelvic nodal radiation in the FASTR-2 study. In addition, given the recent evidence supporting the equivalence of 18 months of hormone therapy, compared to 36 months, it was decided to lengthen the duration of hormone therapy in the FASTR-2 study to 18 months (versus 12 months in the FASTR study).

ELIGIBILITY:
Inclusion Criteria:

* High risk prostate cancer
* Has had multidisciplinary consultation with radiation oncologist and urologist
* Age >70 or refuses standard treatment
* No evidence of extra-prostatic disease on screening bone scan and CT scan (non-contrast CT used for CT simulation acceptable)
* Signed written and voluntary informed consent provided.
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Patients not meeting the eligibility criteria
* Prior pelvic radiotherapy or brachytherapy
* Use of anti-coagulation (low molecular weight heparin or Coumadin)
* History of inflammatory bowel disease, Crohn's disease, diverticulitis or collagen vascular disease (other than rheumatoid arthritis)
* Previous treatment for malignancy (other than basal or squamous cell skin cancer) within 3 years of prostate cancer diagnosis
* patients on androgen deprivation therapy > 2 months prior to study enrolment

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-08 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Genitourinary and Gastrointestinal Toxicity at 1 year | Year 1 of follow-up
  Genitourinary and gastrointestinal toxicity measured at year 1 of follow-up using the Common Toxicity Criteria

SECONDARY OUTCOMES:
Disease Free Survival at 3 years | 1, 2, and 3 years of follow-up
  Defined by absence of clinical relapse and prostatic specific antigen (PSA) failure as per the American Society of Therapeutic Radiation and Oncology (ASTRO) Phoenix definition
Quality of Life | 1, 2, and 3 years of follow-up
  Measured using the Prostate Cancer Radiotherapy questionnaire
Genitourinary and Gastrointestinal Toxicity at 2 years | Year 2 of follow-up
  Genitourinary and gastrointestinal toxicity measured at year 2 of follow-up using the Common Toxicity Criteria
  Safety Issue? (FDAAA) Yes
Genitourinary and gastrointestinal toxicity measured at 3 years | Year 3 of follow-up
  Genitourinary and gastrointestinal toxicity measured at year 3 of follow-up using the Common Toxicity Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Bauman, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

REFERENCES:
- [Derived] Bauman G, Ferguson M, Lock M, Chen J, Ahmad B, Venkatesan VM, Sexton T, D'Souza D, Loblaw A, Warner A, Rodrigues G. A Phase 1/2 Trial of Brief Androgen Suppression and Stereotactic Radiation Therapy (FASTR) for High-Risk Prostate Cancer. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):856-62. doi: 10.1016/j.ijrobp.2015.02.046. Epub 2015 Apr 30. PMID 25936597
- See also: Preliminary Results and Toxicity Analysis — https://pubmed.ncbi.nlm.nih.gov/31681864/